CLINICAL TRIAL: NCT03514732
Title: An Open Label, Single Arm, Exploratory Study to Estimate the Range of Improvement of the Quality of Sleep With NOVANUIT® Triple Action in Subjects With Mild to Moderate Sleep Disorders
Brief Title: Study to Evaluate Improvements of the Quality of Sleep With NOVANUIT® Triple Action in Healthy Volunteers With Sleep Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MELATL07959; U1111-1195-6610 (Other: UTN)
Record Dates: First submitted 2018-04-20; First posted 2018-05-02 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Sleep Disorder (Healthy Volunteers)
MeSH Terms: conditions — Sleep Wake Disorders | interventions — Melatonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Novanuit® Triple Action (Experimental): 2 capsules of Novanuit® Triple Action once daily for 2 weeks, 30 minutes to 1 hour before bedtime.
  Interventions: Drug: MELATONIN (MELATL07959)

INTERVENTIONS:
Drug: MELATONIN (MELATL07959) — Pharmaceutical form:Capsule Route of administration: Oral

SUMMARY:
Primary Objective:

To estimate the range of improvement of NOVANUIT® triple action on sleep quality global score.

Secondary Objectives:

* To estimate the range of improvement of NOVANUIT® triple action on following parameters: time for getting asleep, sleep time, number of nocturnal awakening, number of nightmares, sleep quality (score from 0 to 10), and mean tiredness during the day (score from 0 to 10).
* To estimate persistency of NOVANUIT® triple action effects after end of study product consumption.
* To assess dependency to NOVANUIT® triple action after study product cessation.
* To assess tolerance of NOVANUIT® triple action during the study.

DETAILED DESCRIPTION:
Study participation duration for each participant will be 4 weeks including a 2-week treatment period.

ELIGIBILITY:
Inclusion criteria :

* Healthy men or women volunteers, aged from 20 to 75 years included at the moment of the inclusion visit.
* Subject with Body Mass Index (BMI) between 18.5 and 29.9 kg/m² (limits included).
* Good general health (based on subject interview about his/her medical history and on clinical exam realized by investigator).
* Subject willing to follow diet recommendations in accordance with hygiene and dietary advice defined in the protocol.
* Subject suffering from mild to moderate sleep disorders assessed by Insomnia Severity Index (ISI) questionnaire completed during the selection and presenting a score between 7 and 22 (limits excluded).
* Subject covered by a social security or insurance.

Exclusion criteria:

* Subject having consumed medications for sleep disorders (sleeping pills) during the 6 months previous the inclusion visit and throughout the study duration.
* Subject having consumed dietary supplements for sleep disorders during the 3 months previous to inclusion visit and throughout the study duration.
* Subject presenting history of severe chronic disease (cancer, HIV, renal or hepatic failure, hepatic disorders, inflammatory digestive and known malabsorption diseases, arthritis or chronic respiratory insufficiency, etc.) found to be inconsistent for the study follow up by investigator.
* Subject suffering from a chronic or acute pathology causing sleep disorders.
* Subject consuming products with impact on sleep deterioration at the moment of inclusion visit and throughout the study duration, belong to investigator.
* Subject having undergone general anesthesia during the month previous to inclusion visit.
* Subject suffering from eating disorders (anorexia, bulimia, etc.).
* Subject consuming more than 1.5 packet of tobacco per day (30 cigarettes/day or 27 mg of nicotine/day in electronic cigarette).
* Subject with history of known dependency to drugs or alcohol (consuming more than 3 alcohol units per day). In this study, 1 unit of alcohol is defined as 250 mL of beer, 100 mL of wine or 30 mL of spirits.
* Subject having under the care a child who as constant sleep troubles through the night.
* Subject with irregular working hours (day/night shifts, day/night duties, work trip during the study, etc.).
* Subject taking part in another clinical trial simultaneously and/or in the month previous to inclusion visit and/or being in exclusion period of a previous clinical trial.
* Woman planning to be pregnant soon, actually pregnant or lactating.
* Woman without efficient contraceptive method such as: hormonal contraception (including patch, contraceptive ring, etc.), uterine device or any other mechanic contraceptive method, or condom or diaphragm or spermicide, throughout the duration of the study.
* Subject with sensitivity or known allergy to the product used in the study.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2017-07-05 (Actual); Study Completion 2017-07-05 (Actual)

PRIMARY OUTCOMES:
Comparison of the sleep quality | From baseline to Day 21
  Difference in the average score of sleep quality

SECONDARY OUTCOMES:
Comparison of the average scores of sleep quality | From baseline to Day 28
  Difference in the average score of sleep quality
Comparison of time for getting asleep | From baseline to Day 28
  Difference in the average score of time for getting asleep
Comparison of sleep time | From baseline to Day 28
  Difference in the average score of sleep time
Comparison of number of nocturnal awakening | From baseline to Day 28
  Difference in the average score of number of nocturnal awakening
Comparison of number of nightmares | From baseline to Day 28
  Difference in the average score of number of nightmares
Comparison of awakening quality | From baseline to Day 28
  Difference in the average score of awakening quality
Comparison of mean tiredness | From baseline to Day 28
  Difference in the average score of mean tiredness
Adverse events (AEs) | From baseline to Day 28
  Number of participants with AEs
Dependency questionnaire | At Day 28
  Assessment of product's effects dependency at Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi Administrative Office, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org